CLINICAL TRIAL: NCT05752604
Title: Retrospective and Prospective Evaluation of the Impact of Innovative and Conventional Treatments and of Clinical Variables on the Outcome of Thyroid Cancer
Brief Title: Impact of Conventional Treatments and Clinical Variables on Thyroid Cancer
Acronym: THY-CANC
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 05C212
Record Dates: First submitted 2023-02-17; First posted 2023-03-02 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
DTC has a generally favorable prognosis. The possibility to discriminate between patients with aggressive tumors and those with a more indolent behavior may reduce the need for unnecessary treatments. Aim of this observational study is to evaluate how anamnestic, clinical, and histopathological variables may influence the outcome of the enrolled patients, both regarding morbidity and mortality and in terms of therapeutic choices. The study aims to evaluate the prognostic impact of the therapeutic interventions in terms of efficacy and regarding the appearance of adverse events.

ELIGIBILITY:
Inclusion Criteria:

- thyroid cancer diagnosis

Exclusion Criteria:

* patients unable to sign informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all consecutive patients referred to our tertiary clinical center for thyroid cancer
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2032-03-08 (Estimated); Study Completion 2042-03-08 (Estimated)

PRIMARY OUTCOMES:
Dynamic risk stratification | one year from the primary treatment
  impact of the different variables on the DRS
Dynamic risk stratification | five years from the primary treatment
  impact of the different variables on the DRS
Dynamic risk stratification | ten years from the primary treatment
  impact of the different variables on the DRS
Progression-free survival | one year from the primary treatment
  impact of the different variables on the PFS in patients treated with TKI for advanced thyroid cancer
Progression-free survival | five years from the primary treatment
  impact of the different variables on the PFS in patients treated with TKI for advanced thyroid cancer
Progression-free survival | ten years from the primary treatment
  impact of the different variables on the PFS in patients treated with TKI for advanced thyroid cancer
Overall survival | one year from the primary treatment
  impact of the different variables on the OS in patients treated with TKI for advanced thyroid cancer
Overall survival | five years from the primary treatment
  impact of the different variables on the OS in patients treated with TKI for advanced thyroid cancer
Overall survival | ten years from the primary treatment
  impact of the different variables on the OS in patients treated with TKI for advanced thyroid cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, IRCCS, Milan, Italy